CLINICAL TRIAL: NCT04327908
Title: Cross-cultural Adaptation, Translation and Validation of the German Version of the Toronto Extremity Salvage Score (TESS) and Musculoskeletal Tumor Society (MSTS) for Patients With Bone and Soft Tissue Sarcoma in German Speaking
Brief Title: Translation and Validation of the German Version of the Toronto Extremity Salvage Score (TESS) and Musculoskeletal Tumor Society (MSTS)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Principal Investigator, Dammerer Dietmar, MD, Priv.Doz.Dr. Dietmar Dammerer, MSc PhD, Medical University Innsbruck
Other Study IDs: 1/2020
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionaire TESS and MSTS — answering TESS and MSTS questionnaire

SUMMARY:
The MSTS is an evaluation tool used worldwide to assess physical function in patients with musculoskeletal tumors. The questionnaire has already been successfully translated and validated in Portuguese and Japanese.

Both the TESS and the MSTS have already been used in many studies that examined bone and soft tissue tumors - also in German-speaking populations. So far, however, there is no validated German version of these questionnaires.

The aim of the study at hand is to translate the TESS and the MSTS into German and to validate them for patients with bone and soft tissue tumors / sarcomas.

DETAILED DESCRIPTION:
The most common primary bone tumors include osteosarcoma, Ewing's sarcoma and chondrosarcoma. The main symptom in patients with primary bone tumors is pain that can occur at rest or at night. The physical examination often shows swelling and restricted movement of the joints. Malignant bone tumors require multidisciplinary treatment that focuses on the surgical removal of the tumor. The extremity-preserving procedure contrasts with the amputation. Studies show that the functional result after restoration of the limb is superior to the amputation and that the relapse rate and mortality are comparable in both procedures. The goal of tumor resection is therefore to keep the treatment-related restrictions as low as possible, especially with regard to quality of life, function of the extremity and recurrence-free survival of the patients. The improvement of the functional results and longevity of reconstructive procedures remains a major challenge.

The same applies to the treatment of soft tissue sarcomas. However, early diagnosis is often hampered by atypical symptoms such as soft tissue swelling, painful lesions or no symptoms at all and is reported in the literature with an average period of time until the final diagnosis of 3 to 6 months. En bloc resection is the treatment of choice. Radiation therapy, chemotherapy and isolated hyperthermic limb perfusion can be used depending on tumor histology, degree and extent.

The measurement of the clinical outcome is of great importance. In order to objectify, measure and compare the success or failure of treatment with current literature and other tumor centers and to evaluate the invasive surgical procedures. Questionnaires such as the Toronto Extremity Salvage Score (TESS) and the Musculoskeletal Tumor Society (MSTS) were developed to measure the functional results after surgery and heterogeneity.

The TESS is a valid and disease-specific measure for evaluating functional disorders in patients between 12-85 years of age who are treated surgically for a bone or soft tissue sarcoma of the extremities. The questionnaire measures parameters such as Mobility, independence in everyday life, participation in social life and the pursuit of leisure activities. There is a version for the upper and one for the lower extremity with 30 questions each. Each question is rated on a 1-5 scale, with 5 being the value for normal performance. So far there have been studies to validate the TESS in Portuguese, Danish, Korean and Japanese.

The MSTS is an evaluation tool used worldwide to assess physical function in patients with musculoskeletal tumors. The questionnaire has already been successfully translated and validated in Portuguese and Japanese.

Both the TESS and the MSTS have already been used in many studies that examined bone and soft tissue tumors - also in German-speaking populations. So far, however, there is no validated German version of these questionnaires.

The aim of the study at hand is to translate the TESS and the MSTS into German and to validate them for patients with bone and soft tissue tumors / sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* The questionnaire will be tested on patients who are undergoing extremity-conserving surgery for sarcomas at one of the participating centers as part of the clinical routine. The patients are addressed preoperatively by a member of the study team and during their stay in the clinic whether they participate in the study.

Exclusion Criteria:

* Patients who cannot be treated for extremities and patients who are unable to consent are excluded from the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing a limb-salvage procedere in orthopedic oncology surgeries.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2022-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Validation of psychometric properties of questionnaire MSTS and TESS in German translation | one day
  Patient Reported Outcome Measurements: DASH, HHS, WOMAC, SF12v2 e.g.

SECONDARY OUTCOMES:
Define questionnaires content validité: évaluation of translation quality | one day
  Patient Reported Outcome Measurements: DASH, HHS, WOMAC, SF12v2 e.g.

CONTACTS AND LOCATIONS:
Overall Officials: Dietmar Dammerer, MD, MSc, PhD, Principal Investigator — Medical University of Innsbruck, Dept. Orthopaedics

IPD SHARING:
Plan to Share IPD: No